CLINICAL TRIAL: NCT06550609
Title: Treatment of Bolivian L Braziliensis Mucosal Leishmaniasis with Inhaled Pentamidine Plus Oral Miltefosine
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion Nacional de Dermatologia (Other)
Responsible Party: Principal Investigator, Jaime Soto, Principal Investigator, Fundacion Nacional de Dermatologia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABF-BO-100-10
Record Dates: First submitted 2024-08-08; First posted 2024-08-13 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Mucosal Leishmaniasis
Keywords: Leishmaniasis; Mucosal leishmaniasis; Miltefosine; Pentamidine; Combined therapy
MeSH Terms: conditions — Leishmaniasis, Mucocutaneous; Leishmaniasis | interventions — miltefosine

STUDY DESIGN:
Intervention Model Description: This proof-of-concept phase 2 trial will enroll 20 moderate-to-severe ML patients. The primary endpoint is the cure rate for moderate-severe patients in comparison to literature values for miltefosine alone. If mild ML patients present, up to 10 will also be enrolled. The secondary endpoint is demonstrating that the cure rate for mild disease is 90%-100%.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subjects treated (Experimental): Miltefosine TID for 28 days Inhaled pentamidine 300 mg on days 1,3,5,8,10,12,15,17,19,22
  Interventions: Drug: Miltefosine Oral Capsule

INTERVENTIONS:
Drug: Miltefosine Oral Capsule — Miltefosine 3 pill per day during 28 days AND pentamidine inhaled 300 mg / d during 10 dosis
  Other Names: Pentamidine isethionate inhaled

SUMMARY:
This is a phase 2 study of the combination of inhaled-pentamidine plus oral miltefosine for Bolivian mucosal leishmaniasis.

DETAILED DESCRIPTION:
The 3 major forms of leishmaniasis are visceral, cutaneous, and mucosal disease. Of these, mucosal leishmaniasis (ML) arguably poses the most difficult therapeutic problem. Although visceral disease (VL) occurs in perhaps 300,000 persons a year and is rapidly fatal since TH1 immunity is lacking, visceral disease is well-treated by drugs. Whereras cutaneous disease (CL) is the most prevalent major form occurring in perhaps 1,000,000 persons a year, TH1 Immunity is present and CL self-resolves in 3-18 months.

CL is treated to speed healing of the cutaneous lesion and, for certain species, to try to prevent dissemination of parasites to the oro-nasal mucosa resulting in mucosal leishmaniasis .

Mucosal leishmaniasis (ML) is estimated to occur as a late sequella in approximately 3% of L braziliensis CL. If there are approximately 130,000 cases per year of L braziliensis cutaneous disease, and 3% of these are succeeded by ML, the approximately 4,000 yearly cases of L braziliensis ML makes ML far less common than VL or CL. However, and in spite of more TH1 immunity than cutaneous disease, self-cure of ML is so rare as to be reportable. The patient with ML experiences inexorable erosion of the cartilage of the nose, pharynx, palate, and larynx. ML has been difficult to treat with classical agents (a cure rate of approximately 71%) Thus, of the 3 common forms of leishmaniasis, ML is the form that combines disease severity with poor response to chemotherapy.

Mucosal disease is perhaps the most chemotherapeutically challenging presentation of the leishmaniases. Unlike cutaneous disease, ML results in significant medical morbidity leading to marked psycho-social difficulty, and even mortality. Unlike visceral disease which although mortal quickly responds to therapy, ML is difficult to cure and relapses are common.

Drug combinations are now accepted approaches for many infectious diseases. Since 2 drugs already have the disadvantages of increased cost and potential increased toxicity, use of non-parenteral agents is an important consideration for any proposed combination. As the only recognized oral antileishmanial agent, miltefosine is the drug on which antileishmanial combinations have been based for visceral disease and for cutaneous disease [thermotherapy plus miltefosine: Soto personal communication].

The goal for a miltefosine-based combination for ML would be to raise the ML miltefosine cure rate for "mild" nasal disease to >90% and to raise the miltefosine cure rate for anatomically extensive disease to >58%. Inhaled pentamidine is a non-parenteral agent which in our pilot study was very successful for mild disease (86% cure) but unsuccessful for moderate or severe disease. The combination of oral miltefosine and inhaled pentamidine is a completely non-parenteral regimen that should lead to >90% cure of mild ML disease and could lead to an improved cure rate of moderate-severe disease. Although two drugs will be administered, adverse events should not be additive because miltefosine does not affect the respiratory tract and inhaled pentamidine is minimally absorbed.

This proof-of-concept phase 2 trial will enroll 20 moderate-to-severe ML patients. The primary endpoint is the cure rate for moderate-severe patients in comparison to literature values for miltefosine alone. If mild ML patients present, up to 10 will also be enrolled. The secondary endpoint is demonstrating that the cure rate for mild disease is 90%-100%.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Male or female
* Age: >12 yrs of age
* Weight: > 45 kg
* Consent: Prior to any investigations
* Mucosal disease: Involvement of the nares, nasal mucosa, palate, pharynx, larynx according to the ENT specialist.
* Parasitology: Parasitological confirmation of the lesion (s) will be made by visualization of Leishmania, culture of Leishmania, or molecular identification of Leishmania (PCR) from the biopsy or aspirate of the lesion (s); or a positive Leishmanin skin test plus a scar characteristic of cutaneous leishmaniasis, plus the epidemiologic antecedent of living now or in the past, in an endemic area.

Exclusion Criteria:

* Previous treatment for leishmaniasis: No specific or putatively specific therapy (Sb, pentamidine, amphotericin B, miltefosine, imidazoles, allopurinol) in the last 12 months. Patients may have been previously treated with the agents under investigation---miltefosine, pentamidine---if that treatment ended more than 12 months ago and the disease has not diminished in the last 6 months.
* Other diseases: Concomitant diseases by history that would be likely in the PI's opinion to interact, either positively or negatively, with treatment.
* Laboratory : Values of complete blood count, liver function (AST, ALT, alkaline phosphatase), renal function (creatinine, BUN), pancreatic function (lipase), or uric acid beyond 1.5 x Normal Range and that in the PI's opinion would be clinically meaningful.
* EKG: Clinically significant abnormalities.
* Contraception: Women of childbearing age are required to practice reproductive contraception for 5 months after initiating therapy: abstinence or effective contraception defined as 2 forms of contraception [a barrier method (diaphragm, condom, or cervical cap with spermicidal foam, gel, or cream) plus a 2nd barrier method or hormonal contraceptive or intrauterine device] from day 1 through 5 months post therapy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Efficacy | 25 months
  Clinical Score.Qualification compromise in five places (nose skin, nose mucosa, mouh-palate mucosa, pharynx and larynx usind four signs ( erythema, inflamation, infiltration and ulceration) with this scale: 0= absen5t, 1=mild, 2= moderate and 3= severe. Maximun score: 60

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 6 months
  as Measured by the Number of Adverse Drug Reactions. Physical examination data will be listed at screening and at follow up time points. For laboratory data, the values that are below the lower limit or above the upper limit of the normal reference range will be flagged. Those values or changes in values, which are identified as being clinically significant, will be flagged and summarized separately. For physical examination data, any clinically relevant changes

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clinicas, La Paz, La Paz Department, Bolivia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aronson N, Herwaldt BL, Libman M, Pearson R, Lopez-Velez R, Weina P, Carvalho E, Ephros M, Jeronimo S, Magill A. Diagnosis and Treatment of Leishmaniasis: Clinical Practice Guidelines by the Infectious Diseases Society of America (IDSA) and the American Society of Tropical Medicine and Hygiene (ASTMH). Am J Trop Med Hyg. 2017 Jan 11;96(1):24-45. doi: 10.4269/ajtmh.16-84256. Epub 2016 Dec 7. No abstract available. PMID 27927991
- [Background] Carvalho JP, Silva SN, Freire ML, Alves LL, Souza CSA, Cota G. The cure rate after different treatments for mucosal leishmaniasis in the Americas: A systematic review. PLoS Negl Trop Dis. 2022 Nov 17;16(11):e0010931. doi: 10.1371/journal.pntd.0010931. eCollection 2022 Nov. PMID 36395328
- [Background] Cincura C, de Lima CMF, Machado PRL, Oliveira-Filho J, Glesby MJ, Lessa MM, Carvalho EM. Mucosal leishmaniasis: A Retrospective Study of 327 Cases from an Endemic Area of Leishmania (Viannia) braziliensis. Am J Trop Med Hyg. 2017 Sep;97(3):761-766. doi: 10.4269/ajtmh.16-0349. Epub 2017 Jul 19. PMID 28722607
- [Background] Piccica M, Lagi F, Bartoloni A, Zammarchi L. Efficacy and safety of pentamidine isethionate for tegumentary and visceral human leishmaniasis: a systematic review. J Travel Med. 2021 Aug 27;28(6):taab065. doi: 10.1093/jtm/taab065. PMID 33890115
- [Background] Soto J, Toledo J, Valda L, Balderrama M, Rea I, Parra R, Ardiles J, Soto P, Gomez A, Molleda F, Fuentelsaz C, Anders G, Sindermann H, Engel J, Berman J. Treatment of Bolivian mucosal leishmaniasis with miltefosine. Clin Infect Dis. 2007 Feb 1;44(3):350-6. doi: 10.1086/510588. Epub 2006 Dec 27. PMID 17205440